CLINICAL TRIAL: NCT01967771
Title: A Phase I, Open Label, Randomized, Three Period, Fixed Sequence Crossover Study to Evaluate the Effect of Carbamazepine on Dolutegravir Pharmacokinetics in Healthy Adult Subjects (200901)
Brief Title: Effect of Carbamazepine on Dolutegravir Pharmacokinetics in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 200901
Record Dates: First submitted 2013-10-04; First posted 2013-10-23 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: healthy volunteers; drug interaction; carbamazepine; Dolutegravir; pharmacokinetics
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DTG/CBZ (Experimental): All subjects will be assigned to a single-sequence of three treatment periods without washout. Subjects will receive DTG 50 mg once daily (OD) for 5 days (Period 1), followed by CBZ 100 mg twice daily (BID) for 3 days (days 1-3 of Period 2), CBZ 200 mg BID for 3 days (days 4-6 of Period 2), CBZ 300mg BID for 10 days (days 7-16 of Period 2), followed by DTG 50 mg OD in combination with CBZ 300mg BID for 5 days (Period 3).
  Interventions: Drug: DTG; Drug: CBZ

INTERVENTIONS:
Drug: DTG — DTG will be supplied as 50 mg tablet to be administered orally
Drug: CBZ — CBZ will be supplied as 100 mg and 200 mg extended release tablet to be administered orally

SUMMARY:
This study will be a phase I, open label, three period, fixed sequence crossover study to evaluate the effect of Carbamazepine (CBZ) on the steady-state pharmacokinetics of Dolutegravir (DTG) and on the safety and tolerability of DTG. Subjects will have a screening visit within 30 days prior to the first dose of study drug, three treatment periods, and a follow-up visit 7-14 days after the last dose of study drug. There is no washout between treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including [medical history, physical examination, laboratory tests and cardiac monitoring]. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male/females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, bilateral oophorectomy or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international units per milliliter (MIU/mL) and estradiol <40 picograms (pg)/mL (<147 picomole per liter (pmol/L) is confirmatory]; Child-bearing potential with negative pregnancy test as determined by [serum or urine] human chorionic gonadotropin (hCG) test at screening or prior to dosing AND Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 5 days post-last dose. OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Body weight >=50 kilograms (Kg) for males and >=45 Kg for females and body mass index (BMI) within the range 18.5 - 31.0 Kg/m^2 (square meters) (inclusive).
* Alanine aminotransferase, alkaline phosphatase and bilirubin <= 1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
* Based on single corrected QT interval (QTc) value: QT duration corrected for heart rate by Bazett's formula (QTcB) <450 millisecond (msec); or QTc <480 msec in subjects with Bundle Branch Block.
* A negative HLA-B*1502 allele screening assessment for subjects of Asian ethnicity only.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Pregnant females as determined by positive [serum or urine] hCG test at screening or prior to dosing.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation. Subjects will allergy to tricyclic antidepressants should not be enrolled.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Lactating females.
* The subject's systolic blood pressure is outside the range of 90-140 millimeters of mercury (mmHg), or diastolic pressure is outside the range of 45-90 mmHg, or heart rate is outside the range of 50-100 beats per minute (bpm) for female subjects or 45-100 bpm for male subjects. A single repeat is allowed for eligibility determination.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate for males <45 and >110 bpm and females <50 and >100 bpm; PR interval <120 and >220 msec, QRS duration <70 and >120 msec, QTc interval (Bazett) >450 msec. Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization); any clinically significant arrhythmia which, in the opinion of the investigator and GSK Medical Monitor, will interfere with the safety for the individual subject; any conduction abnormality (including but not specific to left or right incomplete bundle branch block, atrioventricular block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses>3 seconds, and non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).
* Platelets, white blood cell count or hemoglobin below the lower limit of normal. A single repeat is allowed for eligibility determination.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of suicide ideation or severe depression.
* History of hepatic porphyria (e.g., acute intermittent porphyria, variegate porphyria, porphyria cutanea tarda.
* History of previous bone marrow depression (e.g., prior viral or drug related bone marrow depression)
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Unwillingness or inability to follow the procedures outlines in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Steady state plasma DTG pharmacokinetics (PK) parameters | Day 5 and Day 26
  PK parameters will include: Steady state plasma DTG concentration at the end of the dosing interval (Ctau), maximum concentration (Cmax), area under the time-concentration curve over the dosing interval [AUC(0-tau)], apparent clearance following oral dosing (CL/F), terminal phase half life (t1/2), concentration at time zero (C0) and minimum concentration (Cmin)

SECONDARY OUTCOMES:
Change from baseline in 12-lead electrocardiogram (ECG) | Up to 40 days
  Single 12-lead ECGs will be obtained at each timepoint
Change from baseline in vital signs | Up to 40 days
  Vital signs will include systolic and diastolic blood pressure and pulse rate
Number of subjects with adverse events (AEs) | Up to 40 days
  AEs will be assessed throughout the study
Toxicity grading of clinical laboratory tests | Up to 40 days
  Laboratory assessments will include haematology, clinical chemistry and urinalysis parameters

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Song I, Weller S, Patel J, Borland J, Wynne B, Choukour M, Jerva F, Piscitelli S. Effect of carbamazepine on dolutegravir pharmacokinetics and dosing recommendation. Eur J Clin Pharmacol. 2016 Jun;72(6):665-70. doi: 10.1007/s00228-016-2020-6. Epub 2016 Feb 22. PMID 26898568